CLINICAL TRIAL: NCT00556530
Title: Genetic Modifiers of 22q11.2 Deletion Syndrome
Brief Title: Examining Genetic Factors That Affect the Severity of 22q11.2 Deletion Syndrome
Status: Recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital of Philadelphia (Other); University of Geneva, Switzerland (Other); University of Toronto, Centre for Addiction and Mental Health (CAMH) (Unknown); Bambino Gesù Children's Hospital IRCCS (Other); University of California, Los Angeles (Other); Cardiff University (Other); Universidad del Desarrollo (Other); Tel Aviv University (Other); KU Leuven (Other); Maastricht University (Other); The Coriell Institute (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1999-201; R01HL084410 (NIH); R01HL157157 (NIH)
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: DiGeorge Syndrome; 22q11.2 Deletion Syndrome
Keywords: Congenital Heart Defects; Single Nucleotide Polymorphisms; Copy Number Variations; Whole Genome Association Study
MeSH Terms: conditions — DiGeorge Syndrome; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No

SUMMARY:
22q11.2 deletion syndrome is a genetic disorder that can cause heart defects, facial abnormalities, and developmental and learning disabilities. The severity of the disorder can vary widely among people. This study will analyze DNA from people with 22q11.2 deletion syndrome to identify genetic variations that may affect the severity of the disorder.

DETAILED DESCRIPTION:
22q11.2 deletion syndrome is a disorder caused by the deletion of a small piece of chromosome 22. Most people with this disorder are missing a sequence of about 3 million DNA building blocks on chromosome 22 within each cell. This disorder affects many areas of the body. People with 22q11.2 deletion syndrome may have heart defects, immune deficiency, kidney abnormalities, hearing loss, and cleft palate or other facial deformities. Many children experience developmental delays and learning disabilities, and they have an increased risk of developing mental illnesses, including schizophrenia, depression, anxiety, and bipolar disorder. All people with 22q11.2 deletion syndrome are missing the same sequence of DNA, but the severity of this disorder varies widely; some people are diagnosed with multiple health and developmental problems, while others experience very few symptoms. In some people, the symptoms may be so minimal that they are not even aware they have 22q11.2 deletion syndrome. This study will examine genetic material-either from blood or saliva-among people with 22q11.2 deletion syndrome. Participants will attend one study visit and undergo either blood or saliva collection. By analyzing the DNA sequences of participants, the study will aim to identify any genetic variations that may affect the severity of 22q11.2 deletion syndrome.

NOTE: Each clinical site is under the governance of its own Institutional Review Board and discretionary clinicaltrials.gov registration.

ELIGIBILITY:
Inclusion Criteria:

* Has 22q11 deletion of 3 megabases (Mb)

Exclusion Criteria:

* Has 22q11 deletion smaller than 3 Mb or no deletion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with 22q11.2 deletion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07; Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bernice E. Morrow, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, New York, New York, United States